CLINICAL TRIAL: NCT00811629
Title: Soluble Form of the Receptor for Advanced Glycation End Products (sRAGE) Levels in the Pulmonary Edema Fluid and Plasma From ICU Patients With ALI/ARDS and Severe Sepsis : an Observational Prospective Study.
Brief Title: Influence of Acute Respiratory Distress Syndrome (ARDS) and Severe Sepsis on sRAGE Levels in ICU Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0042
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome; Severe Sepsis; Septic Shock; Mechanical Ventilation
Keywords: Receptor for advanced glycation end products (RAGE); Soluble RAGE (sRAGE); Acute Lung Injury (ALI); Acute respiratory distress syndrome (ARDS); Severe sepsis; Septic shock; Alveolar epithelium; Mechanical ventilation; Intensive Care Unit (ICU)
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Sepsis; Shock, Septic

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- control group
  Interventions: Other: sRAGE

INTERVENTIONS:
Other: sRAGE — The purpose of this observational prospective study is to determine wether sRAGE could be used in an ICU setting as a potential diagnostic and prognostic marker during ALI/ARDS, regardless of associated severe sepsis or septic shock

SUMMARY:
sRAGE, the soluble form of the receptor for advanced glycation end products, is a novel marker of alveolar epithelial type I cell injury, but is also involved in acute systemic inflammation. The purpose of this observational prospective study is to determine whether sRAGE could be used in an ICU setting as a potential diagnostic and prognostic marker during ALI/ARDS, regardless of associated severe sepsis or septic shock.

DETAILED DESCRIPTION:
BACKGROUND:

The receptor for advanced glycation end products (RAGE was recently identified as a promising new marker of alveolar type I cell injury. RAGE is a member of the immunoglobulin superfamily that acts as a multiligand receptor and is involved in propagating inflammatory responses. While the precise function of RAGE remains unclear, the elevated levels of RAGE, and its soluble isoform sRAGE, correlate with severity of ALI/ARDS in human and animal studies, and RAGE levels could reflect impaired alveolar fluid clearance. Thus, it is possible that elevated levels of RAGE in ALI/ARDS derive in part from RAGE's role in systemic inflammatory cascades rather than purely from its release from alveolar type I cells.

DESIGN NARRATIVE:

This observational prospective clinical study will describe and compare sRAGE levels in the alveolar edema fluid and in the plasma from ICU patients enrolled within the first 24 hours after onset of ALI/ARDS and/or severe sepsis/septic shock, and from patients under mechanical ventilation (control group). Edema fluid and plasma samples will be collected simultaneously on day 1, day 3, day 6, and day 28 (or at ICU discharge), in order to describe kinetics of evolution of sRAGE levels. Undiluted pulmonary edema fluid samples will be collected in intubated patients only, and blood samples will be gathered from an indwelling arterial catheter. The concentrations of sRAGE will be measured in duplicate by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients under mechanical ventilation
* Patients within the first 24 hours after onset of ALI/ARDS according to the 1994 American-European Consensus Conference (AECC)
* Patients within the first 24 hours after onset of severe sepsis or septic shock according to the 1992 ACCP/SCCM Consensus Conference

Exclusion Criteria:

* Pregnancy
* Acute exacerbation of diabetes
* Dialysis for end-stage kidney disease
* Alzheimer's disease
* Amyloidosis
* Evolutive neoplastic lesion

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Definied population
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
sRAGE levels in the plasma from ICU patients within the first 24 hours after onset of ALI/ARDS or severe sepsis/septic shock | within the first 24 hours

SECONDARY OUTCOMES:
To describe kinetics of evolution of sRAGE levels in ICU patients with ALI/ARDS and severe sepsis/septic shock | in UCU patients

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu JABAUDON, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Jabaudon M, Blondonnet R, Roszyk L, Bouvier D, Audard J, Clairefond G, Fournier M, Marceau G, Dechelotte P, Pereira B, Sapin V, Constantin JM. Soluble Receptor for Advanced Glycation End-Products Predicts Impaired Alveolar Fluid Clearance in Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2015 Jul 15;192(2):191-9. doi: 10.1164/rccm.201501-0020OC. PMID 25932660
- [Derived] Jabaudon M, Futier E, Roszyk L, Chalus E, Guerin R, Petit A, Mrozek S, Perbet S, Cayot-Constantin S, Chartier C, Sapin V, Bazin JE, Constantin JM. Soluble form of the receptor for advanced glycation end products is a marker of acute lung injury but not of severe sepsis in critically ill patients. Crit Care Med. 2011 Mar;39(3):480-8. doi: 10.1097/CCM.0b013e318206b3ca. PMID 21220996